CLINICAL TRIAL: NCT00062582
Title: A 24 Week, Placebo-Controlled, Randomized, Parallel Group Study Comparing Roflumilast 500 mcg Daily vs Placebo on Pulmonary Function and Respiratory Symptoms in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Effect of Roflumilast on Pulmonary Function and Respiratory Symptoms in Patients With Chronic Obstructive Pulmonary Disease (COPD) (BY217/M2-110)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY217/M2-110
Record Dates: First submitted 2003-06-09; First posted 2003-06-10 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD
Keywords: Roflumilast; Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

INTERVENTIONS:
Drug: Roflumilast

SUMMARY:
The aim of the study is to compare the effect of roflumilast and placebo on the lung function in patients with COPD.

ELIGIBILITY:
Main Inclusion Criteria:

* Clinical diagnosis of COPD (Chronic Obstructive Pulmonary Disease)
* Currently stable COPD with no change in COPD treatment in the prior 4 weeks

Main Exclusion Criteria:

* Clinical diagnosis of asthma
* Poorly controlled COPD
* Regular need for daily oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2003-06

PRIMARY OUTCOMES:
pulmonary function.

SECONDARY OUTCOMES:
exacerbation rate
quality of life
symptoms
use of rescue medication
safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (37):
- United States (32):
  - ALTANA Pharma, Cities in Alabama, Alabama
  - ALTANA Pharma, Cities in Arizona, Arizona
  - ALTANA Pharma, Cities in California, California
  - ATLANA Pharma, Cities in Colorado, Colorado
  - ALTANA Pharma, Cities in Conneticut, Connecticut
  - ALTANA Pharma, Cities in Delaware, Delaware
  - ALTANA Pharma, Cities in Florida, Florida
  - ALTANA Pharma, Cities in Georgia, Georgia
  - ALTANA Pharma, Cities in Idaho, Idaho
  - ALTANA Pharma, Cities in Indiana, Indiana
  - ALTANA Pharma, Cities in Iowa, Iowa
  - ALTANA Pharma, Cities in Kansas, Kansas
  - ALTANA Pharma, Cities in Kentucky, Kentucky
  - ALTANA Pharma, Cities in Louisiana, Louisiana
  - ALTANA Pharma, Cities in Maryland, Maryland
  - ALTANA Pharma, Cities in Michigan, Michigan
  - ALTANA Pharma, Cities in Missouri, Missouri
  - ALTANA Pharma, Cities in Nebraska, Nebraska
  - ALTANA Pharma, Cities in Nevada, Nevada
  - ALTANA Pharma, Cities in New Jersey, New Jersey
  - ALTANA Pharma, Cities in New York, New York
  - ALTANA Pharma, Cities in North Carolina, North Carolina
  - ALTANA Pharma, Cities in Ohio, Ohio
  - ALTANA Pharma, Cities in Oregon, Oregon
  - ALTANA Pharma, Cities in Pennsylvania, Pennsylvania
  - ALTANA Pharma, Cities in Rhode Island, Rhode Island
  - ALTANA Pharma, Cities in South Carolina, South Carolina
  - ALTANA Pharma, Cities in Texas, Texas
  - ALTANA Pharma, Cities in Utah, Utah
  - ALTANA Pharma, Cities in Virginia, Virginia
  - ALTANA Pharma, Cities in Washington, Washington
  - ALTANA Pharma, Cities in West Virginia, West Virginia
- ALTANA Pharma, Cities in Argentina, Argentina
- ALTANA Pharma, Cities in Canada, Canada
- ALTANA Pharma, Cities in Colombia, Colombia
- ALTANA Pharma, Cities in Mexico, Mexico
- ALTANA Pharma, Cities in Peru, Peru

REFERENCES:
- See also: BY217-M2-110-RDS-2006-07-27.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4475&filename=BY217-M2-110-RDS-2006-07-27.pdf